CLINICAL TRIAL: NCT04644406
Title: PETRA: PErtuzumab and Trastuzumab Biosimilars Real Life Association for the First Line Treatment of HER2-positive Metastatic Breast Cancer, an Observational Prospective Multicenter Study
Acronym: PETRA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0593
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: HER-2 Positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Efficacy of the Pertuzumab-Trastuzumab combination — The efficacy of the pertuzumab in combination with one of the biosimilars of Trastuzumab will be estimated by measuring the PFS at 6 months after the beginning of the treatment.

SUMMARY:
Currently there are five trastuzumab biosimilars approved by EMA (Ogivri® Mylan , Herzuma® Biogaran, Ontruzant® MSD, Trazimera® Pfizer, and Kanjinti® Amgen) for the treatment of HER2-positive breast cancer. EMA's approvals were obtained on phase I pharmacokinetic equivalence trials and phase III clinical trials based on efficacy primary endpoints in the neoadjuvant setting and on Overall Response Rate in metastatic setting. Safety was a secondary endpoints in these trials.

Phase III pivotal trials compared trastuzumab biosimilars to Herceptin® in combination with chemotherapy in the neoadjuvant setting and in the metastatic setting. The trials were designed before the approval of pertuzumab (in the neoadjuvant and metastatic settings). Thus, there is no available prospective data on the safety and efficacy of trastuzumab biosimilars in combination with pertuzumab.

A biosimilar compound can obtain an extrapolation of its indications to those of the reference biological product since bio-similarity has been demonstrated (ie pharmacokinetic equivalence and clinical studies in the most "sensitive" indications). To date, the use of trastuzumab biosimilar in combination with pertuzumab is allowed, but this combination is not supported by neither scientific evidence nor clinical guidelines.

PETRA aims at evaluate the efficacy and safety of the combination of pertuzumab and a trastuzumab biosimilar in real life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Patients ≥ 18 years-old with non-operable, locally advanced, or metastatic HER-2 positive breast cancer Docetaxel, Paclitaxel or Vinorelbine-based chemotherapy administred in combination with any trastuzumab biosimilar and with pertuzumab for the first-line treatment of the non-operable, locally advanced or metastatic HER-2 positive breast cancer.

WHO Performance status 0-2 Measurable or non-measurable (but radiologically evaluable) disease as per modified Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

Adequate cardia function at baseline defined by a left ventricular ejection fraction of 50% or more within 2 months before treatment start

Adequate baseline organ function, evidenced by the following laboratory results within 2 months before treatment start:

Hemoglobin ≥ 9 g/dL Absolute neutrophil count (ANC) ≥ 1500/mm3 Platelet count ≥ 100,000/mm3 Total bilirubin ≤ 1.5 upper limit of normal (ULN), or total bilirubin ≤ 3.0 × ULN in patients with documented Gilbert's Syndrome.

Glomerular Filtration Rate (GFR) ≥ 30 ml/min according to MDRD formula or CKD-EPI formula or Cockcroft and Gault formula SGOT (AST), SGPT (ALT) and alkaline phosphatase ≤ 5 × ULN Patient's consent to data collection

Exclusion Criteria:

* Prior exposure to trastuzumab in the metastatic setting, patients may have received adjuvant or neoadjuvant trastuzumab and/or pertuzumab with an interval of at least 12 months between completion of the adjuvant or neoadjuvant anti-HER2 therapy and the diagnosis of metastatic breast cancer.

History of allergic reactions attributed to compounds of chemical or biological composition similar to trastuzumab, pertuzumab, or to chemotherapy components Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including known HIV, active hepatitis B and/or hepatitis C infection), symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adults with non-operable, locally advanced or metastatic HER-2 positive breast cancer, treated by chemotherapy in combination with any trastuzumab biosimilar and pertuzumab
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
PFS-R | 6 months after inclusion
  The primary end-point is the 6 months PFS-R. It will be defined as the proportion of included patients who achieve complete response (CR), partial response (PR) or stable disease (SD) at 6 months after the beginning of the treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre de lutte contre le Cancer JEAN PERRIN, CLERMONT-FERRAND, Clermont-Ferrand
  - Hôpital Privé Drome Ardèche, Guilherand-Granges
  - CHU Limoges, Limoges
  - Hospices Civils de LYon, Lyon
  - Hôpital Tenon, AP-HP, Paris
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided